CLINICAL TRIAL: NCT01562665
Title: Epidemiological Study to Describe NSCLC Clinical Management Patterns in MENA
Brief Title: Epidemiological Study to Describe Non Small Cell Lung Cancer Clinical Management Patterns in MENA. Lung-EPICLIN/ Gulf
Acronym: Lung-EPICLIN/G
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OAE-XXX-2011/1
Record Dates: First submitted 2012-02-22; First posted 2012-03-26 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Non Small Cells Lung Cancer
Keywords: All patients with NSCLC attending participating hospitals

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- All Population
- Sample of patients will be invited to complete Quality of Life

SUMMARY:
The overall aim of the study is:

To provide accurate and reliable information regarding NSCLC clinical management across MENA region in order to detect unmet medical needs of this disease in terms of:

* Patient and hospital characteristics.
* Diagnostic and treatment approaches: initial and subsequent.
* Follow-up patterns in clinical management.
* Outcomes: symptoms, death, functionality, quality of life.
* Use of resources and burden on patients and health care systems.

DETAILED DESCRIPTION:
Epidemiological study to describe NSCLC clinical management patterns in MENA

ELIGIBILITY:
Inclusion Criteria:

* Confirmed NSCLC diagnosis (e.g. bronchoscope or FNAB), all stages, men and women, attending the responsible department of treating this type of patients for the first time between November 1st, 2011 and August 30th, 2012 For PRO
* Sub-sample:

  * ability to read and write since they will be asked to participate in the PRO part of the study.
* Selection will not be based on the disease stage of each patient, in order to avoid a selection bias.

Exclusion Criteria:

* According to the study design there will not be any exclusion criteria in order to provide a high validity and to obtain the most accurate real daily practice information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Oncology Institutes
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Use of health resources by collecting data about hospital description and characteristics, Disease Diagnosis Procedures and Therapy information | April 2014(26 Months)

SECONDARY OUTCOMES:
Patient-Reported Outcomes (PRO) through self-administered questionnaires and the patients will be asked to complete them at each evaluation visit(25% of the whole sample) | April 2014(26 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Kakil Rasul, CONSULTANT, Principal Investigator — Hamad Medical Corporation, Doha, Qatar; Ahmed El Khodary, CONSULTANT, Principal Investigator — Kuwait Cancer Centre, Al Sabah Hospital, Kuwait; Norbert Drier, CONSULTANT, Principal Investigator — Zayed Military Hospital, Abu Dhabi, United Arab Emirates; Farid Khalifa, CONSULTANT, Principal Investigator — Salmaniya Medical Complex, Bahrain; Mohamed Jaloudy, CONSULTANT, Principal Investigator — Tawam Hospital ,Alain,Abu Dhabi, United Arab Emirates
Locations (3):
- Research Site, Manama, Bahrain
- Research Site, Doha, Qatar
- Research Site, Alain - AbuAhabi, United Arab Emirates

REFERENCES:
- See also: EpiclinStudy_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=965&filename=EpiclinStudy_Synopsis.pdf